CLINICAL TRIAL: NCT05205460
Title: Effectiveness of a 12-week Telerehabilitation Training in People With Long COVID: A Randomized Controlled Trial
Brief Title: Telerehabilitation in People With Long COVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Chia-Ying Lai, Doctor, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A202105159
Record Dates: First submitted 2022-01-24; First posted 2022-01-25 (Actual); Results first posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-02

CONDITIONS: COVID-19
Keywords: Post-COVID; Telerehabilitation
MeSH Terms: conditions — COVID-19 | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based telerehabilitation (Experimental): After graded exercise testing, the participants will receive a single, individual, face-to-face physical activity promotion counseling session (15-20minutes). Then, the participants will start a home-based telehealth exercise training program (30minutes/session, 3 sessions/week for 12weeks, with a total of 36 sessions) combined with heart rate sensing clothes. Exercise type: brisk walking, jogging, or stationary ergometer exercise.
  Interventions: Device: Home-based telerehabilitation
- Education and self-exercise (Active Comparator): After graded exercise testing, the participants will receive a single, individual, face-to-face physical activity promotion counseling session (15-20minutes).
  Then, the patients will maintain their usual lifestyles for 12 weeks without exercise reminders.
  Interventions: Behavioral: Education and self-exercise

INTERVENTIONS:
Device: Home-based telerehabilitation — A home-based exercise mobile app will be offered combined with the heart rate sensing clothes to each participant in the group of home-based telehealth exercise training program. The mobile app provides auto-feedback of heart rate at each exercise training session through the heart rate sensing clothes and alarm function identifying individuals' appropriate exercise intensity (target heart rate) during their exercise based on their exercise prescription calculated and set up inside the app. After completing each exercise training session, the record of training time and heart rate response is simultaneously uploaded to the cloud system of the medical center through the heart rate sensing clothes. The experienced and well-trained nurse checked the cloud system data to monitor participants' adherence to exercise training. In addition, online communication is enabled using LINE software, which provided a platform for patients and researchers to interact with each other through messaging.
  Arms: Home-based telerehabilitation
Behavioral: Education and self-exercise — The participants will receive a exercise prescription suggestion. Then, they will maintain their usual lifestyles without exercise reminders.
  Arms: Education and self-exercise

SUMMARY:
The aim of our study is to investigate the effectiveness of telerehabilitation in Post-COVID patients.

DETAILED DESCRIPTION:
Decreased exercise capacity, persistent dyspnea and easily fatigue are found in some Post-COVID patients. Telerehabilitation has been developed in cardiac and pulmonary diseases such as coronary artery disease and chronic obstructive pulmonary disease for years with good clinical outcomes. However, little is known about the effectiveness of home-based telerehabilitation among Post-COVID patients. Thus, we want to investigate the effectiveness of telerehabilitation among Post-COVID patients, including cardiorespiratory fitness, physical activity amounts, health related quality of life and sleep quality.

ELIGIBILITY:
Inclusion Criteria:

Individuals who had been diagnosed with COVID-19 positive and whose last PCR test or rapid antigen test was negative with the following criteria:

* aged between 20 to 80 years old
* persistent symptoms at least 4 weeks after recovery from COVID-19 infection, including any of the following symptoms: dyspnea, fatigue, cough, headache, chest tightness, palpitations, loss of smell, anxiety, insomnia, brain fog or joint pain
* able to speak and understand Mandarin
* able to walk including those who need the walking aid
* had mobile phones and could easily access the Internet

Exclusion Criteria:

* a history of chronic obstructive pulmonary disease or other respiratory diseases
* a history of arrhythmia,cancer, end-stage renal disease with dialysis, being diagnosed with mental illness, recent stroke within 6 months
* inability to participate because of comorbid neurological or musculoskeletal conditions that produce moderate to severe physical disability
* need all day oxygen support

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shang-Lin Chiang, PhD, Principal Investigator — Department of Physical Medicine and Rehabilitation, Tri-Service General
Locations (1):
- Tri-service general hospital, Taipei, Neihu, Taiwan

REFERENCES:
- [Derived] Lai CY, Lin CH, Chao TC, Lin CH, Chang CC, Huang CY, Chiang SL. Effectiveness of a 12-week telerehabilitation training in people with long COVID: A randomized controlled trial. Ann Phys Rehabil Med. 2024 Jun;67(5):101853. doi: 10.1016/j.rehab.2024.101853. Epub 2024 Jun 1. PMID 38824899

RESULTS

PARTICIPANT FLOW:
Groups:
- Home-based Telerehabilitation: After graded exercise testing, the participants will receive a single, individual, face-to-face physical activity promotion counseling session (15-20minutes). Then, the participants will start a home-based telehealth exercise training program (30minutes/session, 3 sessions/week for 12weeks, with a total of 36 sessions) combined with heart rate sensing clothes. Exercise type: brisk walking, jogging, or stationary ergometer exercise.
  Home-based telehealth exercise training program: A home-based exercise mobile app will be offered combined with the heart rate sensing clothes to each participant in the group of home-based telehealth exercise training program. The mobile app provides auto-feedback of heart rate at each exercise training session through the heart rate sensing clothes and alarm function identifying individuals' appropriate exercise intensity (target heart rate) during their exercise based on their exercise prescription calculated and set up inside the app. After completing each exercise training session, the record of training time and heart rate response is simultaneously uploaded to the cloud system of the medical center through the heart rate sensing clothes. The experienced and well-trained nurse checked the cloud system data to monitor participants' adherence to exercise training. In addition, online communication is enabled using LINE software, which provided a platform for patients and researchers to interact with each other through messaging.
- Education and Self-exercise: After graded exercise testing, the participants will receive only a single, individual, face-to-face physical activity promotion counseling session (15-20minutes).
  Education and self-exercise: The participants will receive a exercise prescription suggestion. Then, they will maintain their usual lifestyles without exercise reminders.
Period: Overall Study
Arm/Group | Home-based Telerehabilitation | Education and Self-exercise
Started | 91 | 91
Completed | 56 | 66
Not Completed | 35 | 25

BASELINE CHARACTERISTICS:
Groups:
- Education and Self-exercise: After graded exercise testing, the participants will receive a single, individual, face-to-face physical activity promotion counseling session (15-20minutes).
  Then, the patients will maintain their usual lifestyles for 12 weeks without exercise reminders.
  Education and self-exercise: The participants will receive a exercise prescription suggestion. Then, they will maintain their usual lifestyles without exercise reminders.
- Total: Total of all reporting groups
Arm/Group | Home-based Telerehabilitation | Education and Self-exercise | Total
Number analyzed (Participants) | 91 | 91 | 182
Age, Customized [Mean (Standard Deviation); unit: years]
  Age(years) | 38.9 (13.1) | 40.8 (11.5) | 39.9 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 33 | 70
  Male | 54 | 58 | 112
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 91 | 91 | 182
Region of Enrollment [Number; unit: participants]
  Taiwan | 91 | 91 | 182
Duration of post-COVID-19 (weeks) [Mean (Standard Deviation); unit: weeks] | 13.1 (7.5) | 11.5 (5.7) | 12.1 (6.5)
Body mass index (kg/m2) [Mean (Standard Deviation); unit: kg/m2] — BMI is calculated as weight (kg) divided by height squared (m²). Higher values indicate greater body mass, with a BMI ≥ 25 classified as overweight and BMI ≥ 30 as obesity.
  kg/m2 | 23.4 (3.9) | 24.3 (5.2) | 23.9 (4.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in Exercise Capacity: Peak Oxygen Uptake (VO2peak) From Baseline to 12 Weeks
Description: The peak oxygen uptake (VO2peak) is measured by graded exercise testing. A cycling ergometer (MGC Ultima CardiO2) is used for cardiopulmonary testing with a incremental ramp protocol (10-W/min). The test will be terminated until patients complained of physical exhaustion or maximal capacity (respiratory exchange ratio (RER) meets 1.2). The change in VO2 peak was calculated as the value at 12 weeks minus the value at baseline. A higher VO2 peak indicates better exercise capacity.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Home-based Telerehabilitation | Education and Self-exercise
Number analyzed (Participants) | 91 | 91
ml/kg/min | 2.4 (4.4) | 1.7 (4.1)

2. Primary Outcome: Change in Exercise Capacity: Workload (Watt) From Baseline to 12 Weeks
Description: The workload (Watt) is measured by graded exercise testing. A cycling ergometer (MGC Ultima CardiO2) is used for cardiopulmonary testing with a incremental ramp protocol (10-W/min). The test will be terminated until patients complained of physical exhaustion or maximal capacity (respiratory exchange ratio (RER) meets 1.2). The change in workload was calculated as the value at 12 weeks minus the value at baseline. A higher workload indicates better exercise capacity.
Time Frame: baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: watts
Arm/Group | Home-based Telerehabilitation | Education and Self-exercise
Number analyzed (Participants) | 91 | 91
watts | 7.0 (12.1) | 7.3 (13.8)

3. Primary Outcome: Change in Exercise Capacity: Anaerobic Threshold (AT) From Baseline to 12 Weeks
Description: The anaerobic threshold (AT) is measured by graded exercise testing. A cycling ergometer (MGC Ultima CardiO2) is used for cardiopulmonary testing with a incremental ramp protocol (10-W/min). The test will be terminated until patients complained of physical exhaustion or maximal capacity (respiratory exchange ratio (RER) meets 1.2). The change in AT was calculated as the value at 12 weeks minus the value at baseline. A higher AT indicates better exercise capacity and endurance.
Time Frame: baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Home-based Telerehabilitation | Education and Self-exercise
Number analyzed (Participants) | 91 | 91
ml/kg/min | 1.2 (3.4) | 1.0 (3.7)

4. Primary Outcome: Change in Lung Function: Forced Expiratory Volume 1 (FEV1) From Baseline to 12 Weeks
Description: The amount of air exhaled (mL) during the first second during a forced expiratory volume test will be measured by spirometry. The change in FEV₁ was calculated as the value at 12 weeks minus the value at baseline. A higher FEV₁ indicates better lung function.
Time Frame: baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Home-based Telerehabilitation | Education and Self-exercise
Number analyzed (Participants) | 91 | 91
liters | 0.0 (0.3) | 0.0 (0.2)

5. Primary Outcome: Change in Lung Function: Forced Vital Capacity (FVC) From Baseline to 12 Weeks
Description: The total amount of air exhaled (mL) during a forced expiratory volume test will be measured by spirometry. The change in FVC was calculated as the value at 12 weeks minus the value at baseline. A higher FVC indicates better lung function.
Time Frame: baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Home-based Telerehabilitation | Education and Self-exercise
Number analyzed (Participants) | 91 | 91
liters | 0.0 (0.3) | -0.1 (0.3)

6. Primary Outcome: Change in Lung Function: FEV1/FVC % From Baseline to 12 Weeks
Description: The measured FEV1 is divided by the measured FVC. he change in FEV₁/FVC was calculated as the value at 12 weeks minus the value at baseline. A higher FEV₁/FVC ratio generally indicates better lung function, while a lower ratio suggests airflow limitation.
Time Frame: baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of FEV1/FVC
Arm/Group | Home-based Telerehabilitation | Education and Self-exercise
Number analyzed (Participants) | 91 | 91
percentage of FEV1/FVC | -1.2 (10.9) | 0.7 (3.4)

7. Primary Outcome: Change in Ventilation/ Perfusion Abnormalities (VE/VCO2) From Baseline to 12 Weeks
Description: The ventilation/ perfusion abnormalities (VE/VCO2)is measured by graded exercise testing.
  A cycling ergometer (MGC Ultima CardiO2) is used for cardiopulmonary testing with a incremental ramp protocol (10-W/min). The test will be terminated until patients complained of physical exhaustion or maximal capacity (respiratory exchange ratio (RER) meets 1.2).
  The change in VE/VCO2 was calculated as the value at 12 weeks minus the value at baseline. A lower VE/VCO2 ratio indicates better ventilatory efficiency and reduced ventilation/perfusion abnormalities.
Time Frame: baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Home-based Telerehabilitation | Education and Self-exercise
Number analyzed (Participants) | 91 | 91
ratio | -0.1 (1.7) | 0.8 (3.6)

8. Primary Outcome: Change in Left Ventricular Function: O2 Pulse From Baseline to 12 Weeks
Description: O2 Pulse is simply oxygen consumption (in ml) divided by heart rate. It is used as an index of stroke volume.The O2 pulse is measured by graded exercise testing. A cycling ergometer (MGC Ultima CardiO2) is used for cardiopulmonary testing with a incremental ramp protocol (10-W/min). The test will be terminated until patients complained of physical exhaustion or maximal capacity (respiratory exchange ratio (RER) meets 1.2). The change in O₂ pulse was calculated as the value at 12 weeks minus the value at baseline. A higher O₂ pulse indicates improved left ventricular function and greater cardiovascular efficiency.
Time Frame: baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: ml/beats
Arm/Group | Home-based Telerehabilitation | Education and Self-exercise
Number analyzed (Participants) | 91 | 91
ml/beats | 0.5 (1.8) | 0.6 (1.6)

9. Primary Outcome: Change in Heart Rate Recovery From Baseline to 12 Weeks
Description: The heart rate recovery is measured by graded exercise testing, including 1 minute and 2 minute recovery.
  A cycling ergometer (MGC Ultima CardiO2) is used for cardiopulmonary testing with a incremental ramp protocol (10-W/min). The test will be terminated until patients complained of physical exhaustion or maximal capacity (respiratory exchange ratio (RER) meets 1.2). The change in heart rate recovery was calculated as the difference between heart rate recovery at 12 weeks and heart rate recovery at baseline. A decrease of < 12 or 22 beats per minute in 1- or 2-min heart rate recovery, respectively, indicates an elevated risk of mortality. A faster heart rate recovery indicates better cardiovascular fitness and autonomic regulation.
Time Frame: baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: beats
Arm/Group | Home-based Telerehabilitation | Education and Self-exercise
Number analyzed (Participants) | 91 | 91
beats
  1-min HR recovery | 1.1 (5.0) | 1.3 (10.2)
  2-min HR recovery | 2.3 (5.3) | 3.2 (8.3)

10. Secondary Outcome: Change in Physical Activity Amounts: Taiwan Version of the International Physical Activity Questionnaire From Baseline to 12 Weeks
Description: Taiwan version of the International Physical Activity Questionnaire. The overall physical activity (MET-min/week), vigorous intensity physical activity (MET-min/week), moderate intensity physical activity (MET-min/week), walking (MET-min/week) are measured.
Time Frame: baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: MET-min/week
Arm/Group | Education and Self-exercise | Home-based Telerehabilitation
Number analyzed (Participants) | 91 | 91
MET-min/week
  Vigorous PA | -13.6 (1234) | 302.4 (1360)
  Moderate PA | -87.6 (4739) | 103.7 (1189)
  Walking behavior | -1239 (2329) | 406 (1205)
  Total PA | -1341 (2690) | 812 (1643)

11. Secondary Outcome: Change in Confidence Level of Exercise: Questionnaire of Self-Efficacy Items From Baseline to 12 Weeks
Description: Questionnaire of Self-Efficacy Items. A five-item self-efficacy measure designed to measure confidence in one's ability to persist with exercising in various situations was developed. A five-point scale is used to rate each item : 1 indicates "not at all confident", 2 indicates "little confident" , 3 indicates "confident", 4 indicates "very confident", 5 indicates "strongly confident".
Time Frame: baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based Telerehabilitation | Education and Self-exercise
Number analyzed (Participants) | 91 | 91
score on a scale | 1.2 (2.4) | -1.1 (2.5)

12. Secondary Outcome: Change in Health-Related Quality of Life: Taiwan Version of World Health Organization Quality-of-Life Questionnaire From Baseline to 12 Weeks (WHOQOL-BREF)
Description: The Taiwanese version of the WHO Quality of Life-BREF (WHOQOL-BREF) with good validity and reliability includes the globally standardized WHOQOL-BREF with 26 items and an additional two locally developed items, making a total of 28 items. It consists of two single-facet items measuring overall quality of life and general health and four domains, including physical (7 items), psychological (6 items), social (4 items), and environmental (9 items) domains. The two additional items are being respected/accepted facet in the social domain and eating/food facet in the environment domain, respectively. The participants rated all items on a scale of 1-5, with higher scores reflecting a greater quality of life. Domain scores were derived by multiplying the mean of the facet scores within each domain by a scaling factor of 4, resulting in potential domain scores ranging from 4 to 20.
Time Frame: baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based Telerehabilitation | Education and Self-exercise
Number analyzed (Participants) | 91 | 91
score on a scale
  physical domain | 0.5 (1.9) | 0.2 (2.0)
  psychological domain | 0.4 (1.8) | 0.1 (2.7)
  social domain | 0.3 (1.5) | 0.3 (2.4)
  environment domain | 0.2 (1.2) | 0.2 (2.1)

13. Secondary Outcome: Change in Sleep Quality: Pittsburgh Sleep Quality Index (PSQI) From Baseline to 12 Weeks
Description: Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances over a l-month time interval. Nineteen individual items generate seven "component" scores and the sum of scores for these seven components yields one global score. (Scores ranged from 0 to 21, with higher scores indicating poor sleep quality.)
Time Frame: baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based Telerehabilitation | Education and Self-exercise
Number analyzed (Participants) | 91 | 91
score on a scale | 0.9 (2.3) | 0.7 (3.0)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Home-based Telerehabilitation | Education and Self-exercise
All-Cause Mortality (participants affected / at risk) | 0/91 | 0/91
Serious Adverse Events (participants affected / at risk) | 0/91 | 0/91
Other Adverse Events (participants affected / at risk) | 0/91 | 0/91

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-25): https://cdn.clinicaltrials.gov/large-docs/60/NCT05205460/Prot_SAP_000.pdf